CLINICAL TRIAL: NCT00056758
Title: Randomized Phase I Evaluation of Immunization With Highly Conserved HIV-1 Derived Peptides and Influenza Matrix Peptide in HIV-1-Infected Subjects on Highly Active Antiretroviral Therapy (HAART) Using Autologous Dendritic Cells Derived From Adherent Monocytic Precursors
Brief Title: HIV Vaccine Designed for HIV Infected Adults Taking Anti-HIV Drugs
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P01AI043664-04 (NIH); P01AI043664-04 (NIH)
Record Dates: First submitted 2003-03-21; First posted 2003-03-24 (Estimated); Last update posted 2007-08-27 (Estimated); Status verified 2007-08

CONDITIONS: HIV Infections
Keywords: HIV-1; HAART; Therapeutic immunization; HIV Therapeutic Vaccine; Treatment Experienced
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Biological: Autologous Dendritic Cell HIV Vaccination

SUMMARY:
This study will evaluate the safety of and immune responses to a dendritic cell vaccination for HIV-1 infection. The vaccine will be made from a patient's own cells combined with small fragments of HIV-1 (made synthetically in a laboratory). These cells will be administered back to the patient either into a vein (intravenously) or the skin (subcutaneously).

DETAILED DESCRIPTION:
Untreated HIV-1 infection is characterized by progressive immune dysfunction and the development of opportunistic infections and AIDS-associated malignancies. Highly active antiretroviral therapy (HAART) has been successful in suppressing HIV replication and restoring partial immune function. However, HIV-specific immunity remains poor, as evidenced by rapid rebound of HIV-1 RNA following HAART withdrawal. Studies of individuals with acute HIV-1 infection, as well as those who are long-term nonprogressors, have suggested that robust HIV-specific immune responses are associated with control of HIV-1 viremia. Dendritic cells (DCs) are potent antigen presenting cells that may increase HIV-specific immune responses. This protocol will evaluate the use of DCs to help control HIV infection.

Patients will be randomized to receive either intravenous or subcutaneous administration of HIV antigen expressing DCs. Each subject will receive two administrations of mature DCs given 3 weeks apart. Subjects will be followed weekly for 8 weeks, then at Weeks 12, 16, 24, 36, and 48. Two doses of DCs will be evaluated (low dose: 1-3 million cells; high dose: 5-10 million cells) for safety and immune system response.

ELIGIBILITY:
Inclusion Criteria

* HIV-1 infection
* Current CD4 count more than 400/mm3
* HIV RNA less than 400 copies/ml
* Stable combination antiretroviral therapy for at least 4 weeks prior to study entry
* HLA A2.1 (to be tested at screening)

Exclusion criteria

* Prior HIV vaccine
* Systemic steroids or immunosuppressive drugs within 30 days of study entry
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18
Dates: Start 2003-02

PRIMARY OUTCOMES:
Safety and tolerability of peptide pulsed, autologous, cultured dendritic cells

CONTACTS AND LOCATIONS:
Overall Officials: Sharon A. Riddler, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pitt Treatment Evaluation Unit, Pittsburgh, Pennsylvania, United States